CLINICAL TRIAL: NCT07109765
Title: Real-World Evaluation of Secukinumab in Moderate-to-Severe Hidradenitis Suppurativa
Brief Title: Secukinumab Treatment for Moderate to Severe Hidradenitis Suppurativa
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Xiao Ma, Resident physician of dermatology, Peking Union Medical College
Other Study IDs: No. I-24PJ1844
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; Secukinumab; ultrasound
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — secukinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Secukinumab — secukinumab 300 mg weekly for five weeks, followed by 300 mg monthly subcutaneous injection

SUMMARY:
This single-center, prospective, observational study aimed to evaluate the efficacy and safety of Secukinumab in treating moderate-to-severe hidradenitis suppurativa (HS). The study was conducted from June 1, 2025, to June 1, 2026, and all participants were treated at the Department of Dermatology, Peking Union Medical College Hospital. The study was approved by the Clinical and Research Ethics Committee of the Chinese Academy of Medical Sciences, Peking Union Medical College Hospital (Ethics Approval No. I-24PJ1844). All procedures involving human participants adhered to the Declaration of Helsinki. Written informed consent form was signed and obtained from the participant.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* diagnosis of moderate-to-severe HS with Hurley stage II or III
* Disease duration of ≥6 months, presence of at least one draining tunnel or two inflammatory nodules
* inadequate response to prior treatments, such as antibiotics, isotretinoin, or TNF inhibitors

Exclusion Criteria:

* active infections (e.g., viral hepatitis, active tuberculosis)
* use of other biologics or systemic immunosuppressants within the past three months
* severe organ dysfunction (e.g., hepatic or renal failure)
* any other conditions that might affect study results

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants were treated at the Department of Dermatology, Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | From enrollment to the end of treatment at Week 12
  a ≥50% reduction in the combined count of inflammatory nodules and abscesses from baseline, without an increase in the number of abscesses or draining tunnels

SECONDARY OUTCOMES:
Dermatology Life Quality Index | From enrollment to the end of treatment at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- No. 1 Shuai Fu Yuan, Dongcheng District, Beijing, Beijing, Beijing Municipality, China

DOCUMENTS (1):
  • Study Protocol (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT07109765/Prot_000.pdf